CLINICAL TRIAL: NCT01047358
Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Aromasin In The Patients With Early Or Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991089
Record Dates: First submitted 2009-12-24; First posted 2010-01-12 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ajuvant group: adjuvant setting after two to three years of tamoxifen
  Interventions: Drug: Aromasin
- palliative group: palliative setting after progression of disease with anti-estrogen therapy
  Interventions: Drug: Aromasin

INTERVENTIONS:
Drug: Aromasin — 25 mg table QD
  Other Names: exemestane
  Groups: ajuvant group
Drug: Aromasin — 25 mg table QD
  Other Names: exemestane
  Groups: palliative group

SUMMARY:
This non-interventional study is to monitor use in real practice in Korea including adverse events on Aromasin (Exemestane).

DETAILED DESCRIPTION:
All cases at the participating institutions.

ELIGIBILITY:
Inclusion Criteria:

* - Postmenopausal women with breast cancer eligible for hormonal therapy.

Exclusion Criteria:

* Pregnant breast-feeding premenopausal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Postmenopausal women diagnosed as estrogen-receptor positive early breast cancer, who have received two to three years of tamoxifen and are switched to AROMASIN for completion of a total of five consecutive years of adjuvant hormonal therapy OR postmenopausal women with breast cancer that has progressed following anti-estrogen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- South Korea (22):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Myongji Hospital, Kwangdong Unversity College of Medicine, Goyang-si, Gyeonggi-do
  - Wonkwang University School of Medicine and Hospital (WUH), Iksan -si, Jeollabuk-do
  - Asan Medical Center, Seoul, Korea
  - Seoul National University Hospital (SNUH), Seoul, Seoul
  - Hwasun Hospital, Chonnam National University, Cheonnam, South Jeolla Province
  - Inje University Busan Paik Hospital, Busan
  - Yeung Nam University Hospital, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Yonsei Cancer Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, University of Ulsan, Seoul
  - Korea University Medical Center (KUMC) - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991089&StudyName=Post%20Marketing%20Surveillance%20Study%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Aromasin%20In%20The%20Patients%20With%20Early%20Or%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between June 2010 and June 2014 from 25 Korean health care centers.
Groups:
- Aromasin: Participants were included if they had early breast cancer for adjuvant hormonal therapy or advanced breast cancer for second-line hormonal therapy after anti-estrogen therapy and were prescribed Aromasin for the first time. Aromasin was administered as part of routine care. The use and dosage recommendations for aromasin were based on the approved local product document. Any adjustments were made solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Aromasin
Started | 206
Completed | 206 (At least one safety assessment (Safety Population))
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aromasin
Number analyzed (Participants) | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 0
Treatment Indication [Number; unit: Participants]
  Adjuvant Therapy for Early Breast Cancer | 81
  Second-Line Therapy for Advanced Cancer | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: All AEs reported after start of administration of Aromasin were considered as TEAEs and summarized.
Time Frame: From the first dose of Aromasin through the end of the study for an average of 5.6 months
Population: Safety Analysis Set: included participants who received Aromasin at least once and were evaluated upon its related safety endpoints at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aromasin
Number analyzed (Participants) | 206
Percentage of Participants | 25.24

2. Secondary Outcome: Percentage of Participants Without Recurrence/Metastasis (Early Breast Cancer)
Description: The antitumor efficacy for early breast cancer was measured by recurrence/metastasis status (Yes or No) of the participant at the end of the study. The investigator recorded the final evaluation date and the information of tumor recurrence or metastasis (Yes or No) in each participant's case report form (CRF).
Time Frame: At the end of the study, average of 5.6 months.
Population: Efficacy Analysis Set: included all participants who received Aromasin for at least 4 weeks in treatment of breast cancer and had efficacy data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aromasin
Number analyzed (Participants) | 74
Percentage of Participants | 95.95

3. Secondary Outcome: Time-to-Progression (Early Breast Cancer)
Description: Time-to-Progression was defined as the duration from the date of first administration of Aromasin to the date of recurrence or contralateral breast cancer.
Time Frame: At the end of the study, average of 5.6 months
Population: This outcome was planned to be analyzed in participants with early breast cancer in the efficacy analysis set. However, the analysis was not performed because the data of time-to-progression was not captured in the CRF.
Arm/Group | Aromasin
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants by Overall Tumor Response Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) (Advanced Breast Cancer)
Description: The antitumor efficacy for advanced breast cancer was measured by objective tumor assessments according to the RECIST of uni-dimensional evaluation. Complete response (CR) was defined as disappearance of all target and non-target lesions, and no new lesions. Partial response (PR) was defined as disappearance of all target lesions, a persistence of ≥1 non-target lesions, no new lesions; or a ≥30% decrease in the sum of the longest dimensions of the target lesions, no unequivocal progression of existing non-target lesions, no new lesions. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), no unequivocal progression of existing non-target lesions, and no new lesions. PD was defined as a ≥20% increase in the sum of the longest dimensions of the target lesions; or unequivocal progression of existing non-target lesions, or the appearance of ≥1 new lesions.
Time Frame: At the end of the study, average of 5.6 months
Population: Efficacy Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aromasin
Number analyzed (Participants) | 112
Percentage of Participants
  CR | 0.89
  PR | 4.46
  SD | 49.11
  PD | 45.54

ADVERSE EVENTS:
Time Frame: From first dose of Aromasin through the end of the study for an average of 5.6 months.
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Aromasin
Serious Adverse Events (participants affected / at risk) | 2/206
Other Adverse Events (participants affected / at risk) | 40/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aromasin (N=206)
CONDITION AGGRAVATED (General disorders) | 1
ASTHENIA (General disorders) | 1
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aromasin (N=206)
LEG PAIN (General disorders) | 4
OEDEMA PERIPHERAL (General disorders) | 3
HEADACHE (Nervous system disorders) | 5
BILIRUBINAEMIA (Hepatobiliary disorders) | 3
SERUM GLUTAMIC OXALOACETIC TRANSAMINASE INCREASED (Hepatobiliary disorders) | 5
SERUM GLUTAMIC PYRUVIC TRANSAMINASE INCREASED (Hepatobiliary disorders) | 4
PHOSPHATASE ALKALINE INCREASED (Metabolism and nutrition disorders) | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5
SKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
ANOREXIA (Psychiatric disorders) | 3
DEPRESSION (Psychiatric disorders) | 3
INSOMNIA (Psychiatric disorders) | 5
COUGHING (Respiratory, thoracic and mediastinal disorders) | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 3
LYMPHOEDEMA (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days